CLINICAL TRIAL: NCT05545644
Title: : Developing a Brief Family-Involved Treatment for Alcohol Use Disorders
Brief Title: Brief Family-involved Treatment for Alcohol Use Disorder
Acronym: B-FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34AA023304 (NIH)
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: Alcohol Use Disorder
Keywords: alcohol; treatment; brief intervention; family
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Patients randomly assigned, prospectively, to one of two study arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Family-Involved Treatment for Alcohol Use Disorder (B-FIT_ (Experimental): Up to 3 sessions of family-involved treatment for patients with alcohol use disorder (AUD) and a family member: Session 1; psychoeducation; increasing supportive behaviors, enhancing positive activities. Session 2: Improving communication; recovery contracts. Session 3: Review of session1 & 2 interventions; continue with communication skills.
  Interventions: Behavioral: Brief Family-Involved Treatment for Alcohol Use Disorder
- Treatment as Usual (TAU (Active Comparator): Treatment as usual in inpatient AUD rehabilitation program, including daily therapy groups, individual counseling, and health and recreational activities.
  Interventions: Behavioral: Brief Family-Involved Treatment for Alcohol Use Disorder

INTERVENTIONS:
Behavioral: Brief Family-Involved Treatment for Alcohol Use Disorder — Up to 3 sessions of counseling involving a patient with alcohol use disorder and a concerned family member
  Other Names: B-FIT

SUMMARY:
Family-involved treatments for alcohol use disorders (AUDs) hold considerable promise to improve engagement and compliance with treatment and improve treatment outcomes. Currently, however, these treatments are time-intensive and difficult to learn and to integrate with on-going clinical treatment. Consistent with the general trend toward briefer treatments, we propose to develop a brief, 3-session, family-involved treatment that can be incorporated into a variety of other AUD treatment modalities. If successful, the treatment may increase the efficiency and effectiveness of AUD treatment.

DETAILED DESCRIPTION:
The overall aim of this treatment development study is to develop an efficacious, brief, family-involved treatment that can be used flexibly in on-going alcohol treatment settings to advance the dissemination of evidence-based treatment. The treatment to be developed and tested in this grant, "B-FIT" (Brief Family-Involved Treatment), builds on the PI's earlier National Institute on Alcohol Abuse and Alcoholism (NIAAA)-supported efficacy trials and studies of mechanisms of change in Alcohol Behavioral Couple Therapy (ABCT) and is designed as an add-on to community-based substance abuse treatment-as-usual (TAU). B-FIT uses family involvement to enhance patient treatment adherence and outcomes by improving family functioning and increasing family-provided incentives for treatment adherence and abstinence. Study aims are carefully sequenced to develop the B-FIT approach and to judge its merits through a rigorous set of fidelity analyses, a small-scale clinical trial, and prospective tests of potential active ingredients, mediators, and moderators of treatment response. Specific are to: (1) modify ABCT to make it (a) appropriate for any concerned family member, (b) shorter, (c) focused on key mechanisms of change, (d) appropriate for use as part of an on-going alcohol treatment program, and (e) more efficacious by incorporating behavioral contracting procedures; (2) conduct a small-scale clinical trial of B-FIT; and (3) finalize materials for a larger-scale RCT. To accomplish study aims, a stage 1A successive cohort treatment development approach followed by a stage 1B small randomized clinical trial (RCT) will be completed. In the 1A stage, key interventions in B-FIT will be identified and integrated into the preliminary version of the treatment manual. Then, in the 1B stage B-FIT will be tested in an RCT to determine feasibility and preliminary efficacy. The project includes six phases: (1) focus groups with service providers, patients, and concerned family members (CFMs) of patients to obtain feedback about the B-FIT content and materials; (2) modification of the B-FIT protocol in response to the focus group feedback; (3) clinician training in the B-FIT protocol followed by pilot testing with six patients and their CFMs. Each clinician, patient, and CFM will be debriefed after the treatment to assess the B-FIT intervention. (4) Further modifications to the B-FIT materials in response to feedback from the pilot study as well as a second set of focus groups used to obtain feedback on the B-FIT written materials in terms of readability, relevance, and ease of use. (5) Structured didactic and experiential training for clinicians on the B-FIT treatment. (6) A small-scale, randomized clinical trial of TAU versus B-FIT + TAU will be conducted with 60 patients and their CFMs to (a) test the feasibility of B-FIT and impact on patient treatment retention, (b) obtain effect size estimates for pre-post changes in drinking, CFM, and family functioning; (c) assess therapist fidelity; (d) measure hypothesized active ingredients in the treatment; and (e) conduct initial moderator analyses. In parallel with phases 1-5 all measures and study procedures will be finalized. Three-month follow-up data will be collected as part of the clinical trial.

ELIGIBILITY:
Inclusion Criteria, Patient:

* Having a family member rated as important, very important or extremely important
* Score of 8 or higher on the Alcohol Use Disorders Identification Test (AUDIT)
* Negative responses to the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders - 4th edition (DSM-IV) psychotic screener (no to all questions or if any positive symptoms occurred only in the context of substance use)
* Negative responses to a two-question domestic violence screener.

Inclusion Criteria, Family:

* Willing to participate in the study
* AUDIT < 8
* Negative responses to the Structured Clinical Interview for DSM-IV (SCID) psychotic screener
* Negative on a domestic violence screener

Exclusion Criteria, Patient:

* No available important family member
* Score < 8 on AUDIT
* Current psychotic features
* Current domestic violence

Exclusion Criteria, Family:

* Unwilling to participate
* Score of 8 or higher on AUDIT
* Current psychotic features
* Current domestic violence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara S McCrady, PhD, Principal Investigator — University of New Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCrady BS, Tonigan JS, Fink BC, Chavez R, Martinez AD, Borders A, Fokas K, Epstein EE. A randomized pilot trial of brief family-involved treatment for alcohol use disorder: Treatment engagement and outcomes. Psychol Addict Behav. 2023 Nov;37(7):853-862. doi: 10.1037/adb0000912. Epub 2023 Mar 16. PMID 36931829

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a publicly funded inpatient substance use disorder treatment program.
Period: Overall Study
Arm/Group | Brief Family-Involved Treatment for Alcohol Use Disorder (B-FIT_ | Treatment as Usual (TAU
Started | 18 | 17
Completed | 14 | 14
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brief Family-Involved Treatment for Alcohol Use Disorder (B-FIT_ | Treatment as Usual (TAU | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.06 (10.14) | 44.65 (9.49) | 43.31 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 14 | 13 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 7
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 35
Alcohol Use Disorders Identification Test (AUDIT) [Mean (Standard Deviation); unit: units on a scale] — The AUDIT is a 10-item questionnaire designed to screen for alcohol use disorder. It was administered by interview for the current study but can also be used as a self-report measure. Each item is scored on a 0-4 scale, with scores ranging from 0-40. Questions query alcohol use, symptoms of dependence on alcohol, and negative consequences from alcohol consumption. All items are summed to create a total score. A higher score indicates a more severe alcohol use disorder.
  units on a scale | 33.88 (5.12) | 33.53 (5.69) | 33.71 (5.33)
Timeline Followback Interview [Mean (Standard Deviation); unit: Proportion of days abstinent] — The TimeLine FollowBack (TLFB) is an interviewer collected measure, for which the participant reports the number of standard drinks of alcohol consumed on each day during the period of interest. The total number of days on which the participant reports abstinence is counted and divided by the total number of days in the period queried, resulting in the proportion of days abstinent, which can range from 0-1.0.
  Proportion of days abstinent | .35 (.33) | .19 (.31) | .27 (.33)
Family Environment Scale - conflict subscale [Mean (Standard Deviation); unit: Units on a scale] — The Conflict subscale from the Family Environment Scale (FES) measures the amount of openly expressed anger and conflict among family members. This self-report subscale (and the cohesion scale) were the only FES subscales administered. Raw scores are converted to standardized scores based on the FES scoring manual. Standardized scores for the Conflict scale range from 4-65.
  Units on a scale | 5.56 (8.00) | 5.18 (2.16) | 5.37 (1.73)
Family Environment Scale - cohesion subscale [Mean (Standard Deviation); unit: units on a scale] — The Cohesion subscale from the Family Environment Scale (FES) measures the degree of commitment, help, and support family members provide for one another. This self-report subscale (and the conflict scale) were the only FES subscales administered. Raw scores are converted to standardized scores based on the FES scoring manual. Standardized scores for the Cohesion scale range from 33-80.
  units on a scale | 3.61 (1.29) | 3.18 (1.16) | 3.4 (1.22)

OUTCOME MEASURES:

1. Primary Outcome: Form-90 Timeline Followback Interview
Description: The Timeline Followback (TLFB) Interview is one section of a larger interview designed to measures outcomes of alcohol treatment. An interviewer uses a calendar to elicit information from the participant about the amount of alcohol consumed on each day within the time period of interest (3 months prior to the interview at baseline; 4 months from baseline at the follow-up interview). From the daily drinking data on the calendar, the interviewer counts the number of days abstinent, and divides that by the total number of days covered in the interview to generate a single value - proportion of days abstinent. This value can range from 0-100. A family member also was interviewed to provide the same data at follow-up. If follow-up data were unavailable from the participant, the family member report was used. Proportion of days abstinent is the outcome variable of interest. Higher values reflect a more positive outcome.
Time Frame: 120 days
Population: Report of proportion days abstinent based on combined reports of patients and a significant other. Data were not available for 4 participants in the B-FIT condition, and 5 participants in the TAU condition, resulting in a follow-up sample of 14 in B-FIT and 12 in TAU.
Measure: Mean (Standard Deviation); unit: proportion of days abstinent
Arm/Group | Brief Family-Involved Treatment for Alcohol Use Disorder (B-FIT_ | Treatment as Usual (TAU
Number analyzed (Participants) | 14 | 12
proportion of days abstinent | .78 (.06) | .64 (.10)
Statistical Analysis 1: Comparison: Brief Family-Involved Treatment for Alcohol Use Disorder (B-FIT_ vs Treatment as Usual (TAU; Test type: Superiority; Given the small sample size, we relied more heavily on effect size calculations (Hedges g adjusted for small sample bias); Hedges g = .48, Standard Error of Mean .48

2. Secondary Outcome: Drinker Inventory of Consequences (DrInC-2R)
Description: The DrInC-2R is a 45-item self-report of negative consequences of drinking. Respondents report how often each of 45 different potential negative consequences of drinking has occurred, using a 4-point scale ranging from 0 (never) to 3 (almost daily). Higher scores reflect a higher number and frequency of negative consequences. Total scores can range from 0-135.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brief Family-Involved Treatment for Alcohol Use Disorder (B-FIT_ | Treatment as Usual (TAU
Number analyzed (Participants) | 11 | 11
units on a scale | 18.82 (4.76) | 12.71 (4.52)
Statistical Analysis 1: Comparison: Brief Family-Involved Treatment for Alcohol Use Disorder (B-FIT_ vs Treatment as Usual (TAU; Test type: Superiority; [p-value comment as in outcome 1, analysis 1]; Hedges g = .37, Standard Error of Mean .45

3. Secondary Outcome: Family Environment Scale (FES), Conflict Subscale
Description: The Conflict subscale of the FES is a measure the amount of openly expressed anger and conflict among family members. Respondents answer "true" or "false" to each of the nine items on the scale. After the nine items are totaled, the score is converted to a standard score, which ranges from 33-80, based on the norms in the manual. Higher scores indicate more perceived anger and conflict in the family. The Conflict (and Cohesion) were the only FES subscales administered.
Time Frame: 4 months
Population: Participants who completed the measure (11/18 in B-FIT) (11/17 in TAU)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brief Family-Involved Treatment for Alcohol Use Disorder (B-FIT_ | Treatment as Usual (TAU
Number analyzed (Participants) | 11 | 11
units on a scale | 5.45 (.47) | 5.64 (.35)
Statistical Analysis 1: Comparison: Brief Family-Involved Treatment for Alcohol Use Disorder (B-FIT_ vs Treatment as Usual (TAU; Test type: Superiority; [p-value comment as in outcome 1, analysis 1]; Hedges g = .04, Standard Error of Mean .42
Statistical Analysis 2: Comparison: Brief Family-Involved Treatment for Alcohol Use Disorder (B-FIT_; Test type: Superiority — Given the small sample size, we relied more heavily on effect size calculations (Hedges g adjusted for small sample bias); Mean Difference (Final Values) = 0.19; Hedges g = .04; SE = .42

4. Secondary Outcome: Family Environment Scale (FES) - Cohesion Subscale
Description: The Cohesion subscale of the FES is a measure of the respondent's perception of the degree of commitment, help, and support family members provide for one another. Respondents answer "true" or "false" to each of the nine items on the scale. After the nine items are totaled, the score is converted to a standard score, which ranges from 4-65 based on the norms in the manual. Higher scores indicate more perceived cohesion in the family. The Cohesion (and Conflict) subscales were the only subscales from the FES.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brief Family-Involved Treatment for Alcohol Use Disorder (B-FIT_ | Treatment as Usual (TAU
Number analyzed (Participants) | 11 | 11
units on a scale | 2.91 (.37) | 3.45 (.37)
Statistical Analysis 1: Comparison: Brief Family-Involved Treatment for Alcohol Use Disorder (B-FIT_ vs Treatment as Usual (TAU; Test type: Superiority; [p-value comment as in outcome 1, analysis 1]; Hedges g = .44, Standard Error of Mean .63

ADVERSE EVENTS:
Time Frame: 4 months
Description: No adverse events noted
Arm/Group | Brief Family-Involved Treatment for Alcohol Use Disorder (B-FIT_ | Treatment as Usual (TAU
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/18 | 0/17

LIMITATIONS AND CAVEATS:
Difficulties in establishing a site for recruitment, recruitment challenges, scheduling of baseline assessments and treatment sessions with family members, and large numbers of patients at the treatment facility leaving against medical advice, all resulted in a smaller number of participants than planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT05545644/Prot_SAP_000.pdf